CLINICAL TRIAL: NCT03442049
Title: Randomized Controlled Trial of Core Stability Training in Patients With Multiple Sclerosis: Biomechanical and Performance Based Analysis of Gait
Brief Title: Effects of Core Stability Training on Gait in Multiple Sclerosis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Baris Cetin, Research Assisstant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO 14/633
Record Dates: First submitted 2018-01-25; First posted 2018-02-22 (Actual); Last update posted 2018-02-22 (Actual); Status verified 2018-02

CONDITIONS: Multiple Sclerosis; Gait Disorders, Neurologic
Keywords: Multiple Sclerosis; Gait; Spinal Stabilization Exercises; Plantar Pressure Distribution; Rehabilitation
MeSH Terms: conditions — Multiple Sclerosis; Gait Disorders, Neurologic

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Spinal stabilization exercises in addition to home exercise program
  Interventions: Other: Physiotherapy - Study group
- Control Group (Active Comparator): Home exercise program
  Interventions: Other: Physiotherapy - control group

INTERVENTIONS:
Other: Physiotherapy - Study group — Study group : In addition to home program spinal stabilization exercises
  Arms: Study group
Other: Physiotherapy - control group — Home exercise program
  Arms: Control Group

SUMMARY:
Gait and mobility are among the functions frequently affected in Multiple Sclerosis (MS) and have a negative impact on quality of life. Strength losses in lower limb muscles, ataxia, sensory problems and fatigue are the most important reasons of walking problems in patients with MS. In addition to loss of strength and tonus problems, especially biomechanical disorders can be seen on foot and this problem affects gatin and balance negatively. The stabilizing muscles, defined as the "core" region and enveloping the body like a corset, are active in the context of postural preparation prior to lower extremity movements and stabilize for the limb movements to be performed. The aim of this study was to investigate the effects of spinal stabilization exercises on walking performance, fatigue, plantar pressure distribution, balance, muscle strength and quality of life in patients with Multiple Sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years old
* EDSS score is between 3-5,5
* Patients who did not take corticosteroid therapy within three months
* Patients who get at least 24 points from the Mini Mental Test were included in the study.

Exclusion Criteria:

* Patients who had an acute MS attack or had an attack within the last three months.
* An orthopedic or systemic problem that would prevent participation in exercises
* Patients who were using walking orthoses or walking aids were not included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-02-20 (Actual); Study Completion 2016-05-01 (Actual)

PRIMARY OUTCOMES:
6 Minutes Walk Test | Change from Baseline 6 Minutes Walking Distance at 6 weeks.
  Maximum Walking Distance in 6 Minutes
Modified Borg Scale | Change from Baseline Fatigue Score at 6 weeks.
  Evaluating fatigue between the scores of 0 and 10. "0" means no fatigue at all. "10" means maximal fatigue.
Plantar Pressure Distribution | Change from baseline peak pressure and contact area values at 6 weeks
  Peak pressure values of 10 subregions under the foot
Plantar Pressure Distribution | Change from baseline peak pressure and contact area values at 6 weeks
  Contact area values of 10 subregions under the foot
Multiple Sclerosis Quality of Life Scale | Change from baseline mental and physical quality of life scores at 6 weeks
  Quality of life assessment with 54 questions about mental and physical health in daily life activities.

SECONDARY OUTCOMES:
Muscle strength with hand held dynamometer | Change from baseline muscle strength at 6 weeks
  Hip Flexors Muscle Strength
Muscle strength with hand held dynamometer | Change from baseline muscle strength at 6 weeks
  Hip Abductors Muscle Strength
Muscle strength with hand held dynamometer | Change from baseline muscle strength at 6 weeks
  Knee Flexors Muscle Strength
Muscle strength with hand held dynamometer | Change from baseline muscle strength at 6 weeks
  Knee Extensors Muscle Strength
Muscle strength with hand held dynamometer | Change from baseline muscle strength at 6 weeks
  Ankle Dorsiflexors Muscle Strength
MiniBESTest | Change from baseline MiniBESTest scores at 6 weeks
  Static and dynamic balance evaluation. This test includes 14 items and maximum score is 28. 28 points means best balance status.
Dynamic Gait Index | Change from baseline Dynamic Gait Index scores at 6 weeks
  Dynamic balance evaluation especially walking balance. This test includes 8 items and maximum score is 24. Maximum score means best dynamic balance status.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bethoux F. Gait disorders in multiple sclerosis. Continuum (Minneap Minn). 2013 Aug;19(4 Multiple Sclerosis):1007-22. doi: 10.1212/01.CON.0000433286.92596.d5. PMID 23917098
- [Background] Givon U, Zeilig G, Achiron A. Gait analysis in multiple sclerosis: characterization of temporal-spatial parameters using GAITRite functional ambulation system. Gait Posture. 2009 Jan;29(1):138-42. doi: 10.1016/j.gaitpost.2008.07.011. Epub 2008 Oct 31. PMID 18951800
- [Background] Freeman JA, Gear M, Pauli A, Cowan P, Finnigan C, Hunter H, Mobberley C, Nock A, Sims R, Thain J. The effect of core stability training on balance and mobility in ambulant individuals with multiple sclerosis: a multi-centre series of single case studies. Mult Scler. 2010 Nov;16(11):1377-84. doi: 10.1177/1352458510378126. Epub 2010 Aug 10. PMID 20699285
- [Background] Hides J, Wilson S, Stanton W, McMahon S, Keto H, McMahon K, Bryant M, Richardson C. An MRI investigation into the function of the transversus abdominis muscle during "drawing-in" of the abdominal wall. Spine (Phila Pa 1976). 2006 Mar 15;31(6):E175-8. doi: 10.1097/01.brs.0000202740.86338.df. PMID 16540858
- [Background] Freeman J, Fox E, Gear M, Hough A. Pilates based core stability training in ambulant individuals with multiple sclerosis: protocol for a multi-centre randomised controlled trial. BMC Neurol. 2012 Apr 5;12:19. doi: 10.1186/1471-2377-12-19. PMID 22480437